CLINICAL TRIAL: NCT01403636
Title: A Phase 2 Study of SAR245409 in Patients With Relapsed or Refractory Mantle Cell Lymphoma, Follicular Lymphoma, Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma or Diffuse Large B Cell Lymphoma
Brief Title: A Study of Investigational SAR245409 in Patients With Certain Lymphoma or Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD12130; 2011-001616-57 (EudraCT Number); U1111-1118-6417 (Other: UTN)
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — XL765

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- mantle cell (Experimental): 50 mg twice daily: no eating for 2 hours prior and 1 hour after dose
  Interventions: Drug: SAR245409
- follicular lymphoma (Experimental): 50 mg twice daily: no eating for 2 hours prior and 1 hour after dose
  Interventions: Drug: SAR245409
- CLL/SLL (Experimental): 50 mg twice daily:no eating for 2 hours prior and 1 hour after dose
  Interventions: Drug: SAR245409
- Diffuse large B cell lymphoma (Experimental): 50 mg twice daily:no eating for 2 hours prior and 1 hour after dose
  Interventions: Drug: SAR245409

INTERVENTIONS:
Drug: SAR245409 — Pharmaceutical form:capsule Route of administration: oral

SUMMARY:
Primary Objective:

- To evaluate the efficacy of SAR245409 as determined by the objective response rate (ORR) in patients with 1 of following relapsed or refractory lymphoma or leukemia subtypes: mantle cell lymphoma (MCL), follicular lymphoma (FL), chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), or diffuse large B cell lymphoma (DLBCL)

Secondary Objectives:

* To assess duration of response, progression free survival (PFS), and proportion of patients with PFS at 6 months (24 weeks) in patients with either MCL, FL, CLL/SLL or DLBCL treated with SAR245409
* To evaluate the safety and tolerability of SAR245409 in patients with MCL, FL, CLL/SLL or DLBCL
* To further characterize the plasma pharmacokinetics (PK) of SAR245409 in patients with MCL, FL, CLL/SLL or DLBCL

DETAILED DESCRIPTION:
There is a 21 day screening period followed by 28 day cycles. Patients will continue to receive SAR245409 as long as there is clinical benefit or until a study withdrawal criterion is met. The last posttreatment visit will be 30 days after the last dose or until IMP-related toxicities have resolved or are deemed irreversible, whichever is later.

ELIGIBILITY:
Inclusion criteria:

* Tissue from an archived or fresh tumor sample
* A peripheral blood buffy coat sample is required for CLL/SLL.
* Patient has mantle cell lymphoma (MCL), follicular lymphoma (FL), or chronic lymphocytic leukemia (CLL)/SLL or diffuse large B cell lymphoma
* Patient > or = 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status < or = 2. Patients with DLBCL will have ECOG < or = 1
* Adequate white blood cells and hemoglobin
* Good kidney and liver function
* Fasting glucose < 160 mg/dL
* No other malignancy
* Use of adequate birth control

Exclusion criteria:

* Treatment with cytotoxic chemotherapy, biologic agents, investigational therapies within 4 weeks, or nitrosoureas or mitomycin C within 6 weeks of study enrollment
* Treatment with a small-molecule kinase inhibitor within 2 weeks, or 5 half lives of the drug or its active metabolites (whichever is longer) of study enrollment
* Prior treatment with a PI3K, mTOR, or Akt inhibitor. Prior treatment of MCL with temsirolimus is permitted in patients enrolled from countries where it is licensed for this indication.
* Radiation therapy within 2 weeks of enrollment
* Autologous stem cell transplantation within 16 weeks of enrollment
* Prior allogeneic transplantation except for patients with R/R DLBCL who meet inclusion criteria
* Central nervous system (CNS) or leptomeningeal involvement. Patients with DLBCL may have active CNS or leptomeningeal involvement.
* Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (anti-HCV) serology
* Primary CNS lymphoma
* Primary mediastinal B-lymphoma

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) as defined as the proportion of patients who experience complete response/remission (CR) or partial response/remission (PR) | 2 months to 2 years

SECONDARY OUTCOMES:
Progression free survival (PFS) at 6 months | 6 months to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (30):
- United States (12):
  - Investigational Site Number 840012, Los Angeles, California
  - Investigational Site Number 840104, Fort Meyers, Florida
  - Investigational Site Number 840006, Augusta, Georgia
  - Investigational Site Number 840011, Maywood, Illinois
  - Investigational Site Number 840010, Kansas City, Kansas
  - Investigational Site Number 840013, Lexington, Kentucky
  - Investigational Site Number 840007, Paducah, Kentucky
  - Investigational Site Number 840004, Boston, Massachusetts
  - Investigational Site Number 840015, St Louis, Missouri
  - Investigational Site Number 840014, Canton, Ohio
  - Investigational Site Number 840001, Philadelphia, Pennsylvania
  - Investigational Site Number 840002, Morgantown, West Virginia
- Australia (4):
  - Investigational Site Number 036002, Clayton
  - Investigational Site Number 036001, Hobart
  - Investigational Site Number 036005, Kingswood
  - Investigational Site Number 036003, Perth
- Belgium (3):
  - Investigational Site Number 056003, Brussels
  - Investigational Site Number 056002, Ghent
  - Investigational Site Number 056001, Leuven
- France (5):
  - Investigational Site Number 250002, Montpellier
  - Investigational Site Number 250001, Pierre-Bénite
  - Investigational Site Number 250004, Rennes
  - Investigational Site Number 250005, Rouen
  - Investigational Site Number 250003, Villejuif
- Germany (3):
  - Investigational Site Number 276003, Frankfurt am Main
  - Investigational Site Number 276002, Jena
  - Investigational Site Number 276001, Ulm
- Netherlands (3):
  - Investigational Site Number 528001, Amsterdam
  - Investigational Site Number 528003, Groningen
  - Investigational Site Number 528002, Rotterdam

REFERENCES:
- [Derived] Brown JR, Hamadani M, Hayslip J, Janssens A, Wagner-Johnston N, Ottmann O, Arnason J, Tilly H, Millenson M, Offner F, Gabrail NY, Ganguly S, Ailawadhi S, Kasar S, Kater AP, Doorduijn JK, Gao L, Lager JJ, Wu B, Egile C, Kersten MJ. Voxtalisib (XL765) in patients with relapsed or refractory non-Hodgkin lymphoma or chronic lymphocytic leukaemia: an open-label, phase 2 trial. Lancet Haematol. 2018 Apr;5(4):e170-e180. doi: 10.1016/S2352-3026(18)30030-9. Epub 2018 Mar 14. PMID 29550382